CLINICAL TRIAL: NCT04622475
Title: Investigator-initiated Trial to Explore the Efficacy and Safety of Fecal Microbiota Transplant (FMT) Capsule in the Treatment of Steroid-refractory Gastrointestinal Acute Graft Versus Host Disease Patients
Brief Title: Efficacy and Safety of FMT Capsule Treating Steroid-refractory GI-aGvHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XBI-302CT1004
Record Dates: First submitted 2020-10-28; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Steroid-refractory Gastrointestinal Acute Graft Versus Host Disease
MeSH Terms: interventions — Fecal Microbiota Transplantation; Capsules

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Fecal Microbiota Transplant (FMT) Capsule
  Interventions: Biological: Fecal Microbiota Transplant (FMT) Capsule

INTERVENTIONS:
Biological: Fecal Microbiota Transplant (FMT) Capsule — When enrolled in the study, subjects will ingest 20 FMT capsules/day orally for 3 consecutive days. If the syndrome is not completely recovered or relapse 14 days after the first administration, the subject will receive a booster dose (20 capsules/day for 3 consecutive days).

SUMMARY:
Gastro-Intestinal Acute Graft Versus Host Disease (GI-aGVHD) is a complication of allogeneic stem cell transplant which is usually treated with steroids. When aGVHD does not respond to steroids it is described as steroid-refractory aGVHD. There is no standard therapy for steroid-refractory GI-aGVHD.

Fecal Microbiota Transplantation (FMT) is the transfer of fecal material from a healthy donor to a patient in order to restore the diversity of the intestinal microbiota. FMT is currently indicated for the treatment of recurrent Clostridium Difficile infection.

The investigators hypothesize that perturbations in the intestinal microbiota following allogeneic hematopoietic stem cell transplantation (HSCT) are essential for the development and propagation of acute graft-versus-host disease. Therefore, modification of HSCT recipients' gut microbiota using fecal transplantation from a healthy donor could be used to treat gut acute GVHD.

This study evaluates safety and feasibility of fecal microbiota transplantation with frozen capsules from healthy donors for the treatment of steroid resistant or steroid dependent acute graft-versus-host disease of the gut.

DETAILED DESCRIPTION:
This trial is designed to reconstruct the intestinal micro-ecology of patients with steroid-refractory gastrointestinal acute graft versus host disease (GI-aGvHD) by FMT. The primary objective is to evaluate the safety of FMT capsule in the treatment of steroid-refractory GI-aGvHD patients. The secondary objectives are as follows.

To observe the efficacy of FMT capsule in the treatment of steroid-refractory GI-aGvHD 28 days after the first administration.

To explore the characteristics of gut microbiota changes after FMT capsule treating steroid-refractory GI-aGvHD.

To evaluate the safety of FMT capsule treating steroid-refractory GI-aGvHD 12 weeks and 24 weeks after the first administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be willing and able to sign the informed consent form and complete the follow-up visits.
2. 18-75 years old. No gender limitation.
3. Patients who can swallow the capsules without chewing.
4. Patients who were clinically diagnosed as steroid refractory GI-aGvHD. The diagnosis criteria are: experiencing GI-aGvHD clinical manifestations (e.g., abdominal cramps, diarrhea, stool blood) within 100 days after receiving hematopoietic stem cell transplant (HSCT); having Grade 2-4 gastrointestinal clinical symptoms; excluding diarrhea caused solely by pathogen infection; after adequate steroid treatment, disease progression on day 3, or with no change on day 7, or without complete response on day 14.
5. Patients who had complicated infection after the diagnosis of aGvHD, but are able to discontinue all the antibiotic therapy 12 hours before receiving FMT treatment.
6. ECOG scale ≤3
7. Basic body function indexes reach the following criteria: total neutrophil≥0.5*10^9/L, platelet count≥100*10^9/L, serum creatinine ≤1.5×upper limit of normal (ULN) or creatinine clearance≥40 mL/min, albumin≥25g/L.

Exclusion Criteria:

1. Patients with extremely serious grade IV aGvHD (life-threatening or with serious non-GvHD complication).
2. Refractory malignant condition.
3. Patients who have received two or more HSCT.
4. Patients who have active infection that has not been controlled and must receive antibiotic therapy, including diarrhea (non-GvHD diarrhea) caused by infection or antibiotics, excluding GvHD complicated infective diarrhea.
5. Patients who have gastrointestinal perforation or toxic intestinal.
6. Patients who have a history of severe allergic reactions.
7. Any condition in which PI do not consider it appropriate to participate (e.g., any medical history, treatment history, or abnormal history of testing data that may confuse the study results, or interfere with the patient's full participation in the study, or hurt the patient's benefit)
8. Female patients who have positive pregnancy test results or are breastfeeding. Women of childbearing age who refuse to use contraception one month after FMT treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The number of adverse events (AEs)/serious adverse events (SAEs) | 28 days
  The number of FMT capsule associated AEs/SAEs occurring from the first administration of FMT to Day 28 (Day 1 is the last day of the first dose of FMT).
The severity of AEs/SAEs | 28 days
  The severity of FMT capsule associated AEs/SAEs occurring from the first administration of FMT to Day 28 (Day 1 is the last day of the first dose of FMT).

SECONDARY OUTCOMES:
Response rate | 28 days
  GI-aGvHD response rate (Complete response+Partial response) on Day 28 after the first dose of FMT (Day 1 is the last day of the first dose of FMT).
Changes in gut microbiota | Days 28, 43, 84, and 168
  Compare the gut microbiota diversity and major bacterial genus before and 28, 43(for subjects recieved 2 dose of FMT), 84 and 168 days after FMT treatment.
The number of AEs/SAEs | Weeks 12 and 24
  The number of FMT capsule associated AEs/SAEs occurring from the first FMT treatment to Weeks 12 and 24 after the first FMT treatment.
The severity of AEs/SAEs | Weeks 12 and 24
  The severity of FMT capsule associated AEs/SAEs occurring from the first FMT treatment to Weeks 12 and 24 after the first FMT treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China